CLINICAL TRIAL: NCT05040698
Title: An Exploratory, Proof-of-Concept Study of the Effect of Fostamatinib Upon Cutaneous Inflammation in the Setting of Hidradenitis Suppurativa
Brief Title: Study of the Effect of Fostamatinib Upon Cutaneous Inflammation in the Setting of Hidradenitis Suppurativa
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Holdsworth House Medical Practice (Other)
Collaborators: Rigel Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, John Frew, Principal Investigator, Holdsworth House Medical Practice
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JFR-001
Record Dates: First submitted 2021-08-30; First posted 2021-09-10 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Hidradenitis Suppurativa
Keywords: fostamatinib; HS; Tavalisse
MeSH Terms: conditions — Hidradenitis Suppurativa | interventions — fostamatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Open Label Fostamatinib (Experimental): Open label Fostamatinib 100mg dose adjusted by the Principal Investigator after week 1
  Interventions: Drug: Fostamatinib

INTERVENTIONS:
Drug: Fostamatinib — Open label Fostamatinib
  Other Names: Tavalisse; R935788

SUMMARY:
A 16 week exploratory, Proof of Concept study to evaluate the effect of Fostamatinib (12 weeks of treatment) upon cutaneous inflammation in Hidradenitis Suppurativa.

DETAILED DESCRIPTION:
Sample size: 20 patients Study duration: 16 weeks

Primary Endpoints:

Alterations in Gene Expression Profiling, cell counts (CD3+, CD11c+, Neutrophil Elastase+, CD20+, CD138+) at Week 4 compared to Baseline.

Alterations in Gene Expression Profiling, cell counts (CD3+, CD11c+, Neutrophil Elastase+, CD20+, CD138+) at Week 12 compared to Baseline.

Secondary Endpoints:

Safety and Tolerability (Grade 2/3 Adverse Effects); Changes in Disease Activity (Measures by AN count and IHS4 scoring).

Study procedures Clinical Examination, Patient Questionnaires, Skin Biopsy, Blood Draw, medical photography

ELIGIBILITY:
Inclusion Criteria:

* Moderate to Severe (Hurley Stage 2 or 3) Hidradenitis Suppurativa as determined by the PI

Exclusion Criteria:

* Uncontrolled hypertension (systolic blood pressure [BP] ≥135 mmHg and/or diastolic BP ≥85 mmHg), unstable angina, congestive heart failure of New York Heart Association classification III or IV, serious cardiac arrhythmia requiring treatment (exceptions: atrial fibrillation, paroxysmal supraventricular tachycardia) at screening.
* History of myocardial infarction within 3 months prior to screening.
* Shock or hypotension requiring vasoactive peptides, such as dopamine, norepinephrine, epinephrine, or dobutamine at screening or at randomization.
* Renal function impairment with creatinine clearance <30 mL/min at screening (estimated glomerular filtration rate will be calculated using the modification of diet in renal disease equation).
* Liver function impairment with aspartate aminotransferase/alanine aminotransferase >=3x the upper limit of normal or bilirubin >2X the upper limit of normal at screening.
* Neutrophil count <1000/µL at screening.
* History of an allergic reaction or hypersensitivity to the study treatment or any component of the study treatment formulation.
* Has documented HIV infection or documented, active hepatitis B or hepatitis C infection.
* Women lactating, pregnant or of childbearing potential who are not willing to avoid becoming pregnant during the study.
* Individuals with concurrent use of systemic antibiotics/ oral retinoids/ systemic immunosuppressants (those with prior use of these medications must have conducted a washout period of 4 weeks or 5 half-lives of the drug, whichever is longer).
* Any medical, psychological or social condition that, in the opinion of the Investigator, would jeopardize the health or well-being of the participant during any study procedures or the integrity of the data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2023-01-13 (Actual); Study Completion 2023-01-27 (Actual)

PRIMARY OUTCOMES:
Week 4 evaluation | 4 weeks
  Alterations in Gene Expression Profiling, cell counts (CD3+, CD11c+, Neutrophil Elastase+, CD20+, CD138+) at Week 4 compared to
Week 12 evaluation | 12 weeks
  Alterations in Gene Expression Profiling, cell counts (CD3+, CD11c+, Neutrophil Elastase+, CD20+, CD138+) at Week 12 compared to Baseline

SECONDARY OUTCOMES:
Grade 2/3 Adverse Events | 12 weeks
  Number of Grade 2/3 Adverse Effects of Fostamatinib over the 12 Week course of treatment.
Abscess and Nodule Count Week 4 | 4 weeks
  Changes in Abscess and Nodule count at Week 4 compared to baseline
International Hidradenitis Suppurativa Severity Score (IHS4) Week 4 | 4 weeks
  Changes in IHS4 score at Week 4 compared to baseline
Abscess and Nodule count week 12 | 12 weeks
  Changes in Abscess and Nodule count at Week 12 compared to baseline
International Hidradenitis Suppurativa Severity Score (IHS4) Week 12 | 12 weeks
  Changes in IHS4 score at Week 12 compared to baseline
Physician Rated Overall Disease Severity | 12 weeks
  Changes in physician rated overall disease severity by visual analogue scale (0-10) at week 12 compared to baseline
Dermatology Life Quality Index (DLQI) | 12 weeks
  Changes in the DLQI (0-30) at week 12 compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: John Frew, MBBS, Principal Investigator — Holdsworth House Medical Practice
Locations (1):
- Holdsworth House Medical Practice, Sydney, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No